CLINICAL TRIAL: NCT06552598
Title: Phase I/II Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Local Administration of Recombinant Oncolytic Adenovirus Injection (KD01) in Patients With Gynecologic Malignancies
Brief Title: The Safety, Tolerability, and Efficacy of KD01 in Gynecologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-TJ-KD01
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Gynecologic Malignancies; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD01 treatment (Experimental): Local administration of Recombinant Oncolytic Adenovirus Injection (KD01) in gynecologic malignancies.
  Interventions: Drug: KD01(the recombinant oncolytic adenovirus)

INTERVENTIONS:
Drug: KD01(the recombinant oncolytic adenovirus) — Drug:
  Phase I: KD01(1×10¹¹ VP, 1×10¹¹ VP, and 6×10¹¹ VP) Phase II Cohort A: KD01(3×10¹¹ VP)+AK104(6 mg/kg)+thymalfasin + rhGM-CSF Phase II Cohort B: KD01(1×10¹¹ VP) + LNG-IUS Administration： Phase I: KD01 will be administered of Cycle 1 (Days 1-5). And subsequent cycles will be repeated every 26 + 7 days thereafter.
  Phase II Cohort A: KD01 will be administered daily on Days 1-5).AK104will be administered on Day 14.KD01 will be resumed daily for up to 5 doses.A second dose of AK104 will be administered on Day 28.Concurrent administration of thymalfasin and rhGM-CSF.Efficacy assessment will be performed on Day 42 . The first elective surgery will be scheduled after evaluation by the investigator.
  Phase II Cohort B: Hysteroscopy will be performed on Day 1; subsequently, KD01 will be administered, and a LNG-IUS will be placed. Thereafter, hysteroscopic diagnostic curettage/biopsy will be carried out every 3 months, accompanied by administration of KD01 and placement of LNG-IUS.

SUMMARY:
Recombinant oncolytic adenovirus injection (KD01)is an oncolytic vius product. Its main component is a conditionally replicativerecombinant human type 5 adenovirus, where part of the E3 region has been replaced with the gene encoding the tBid apoptoticprotein.AK104 is a humanized bispecific antibody co-targeting PD-1 (Programmed Cell Death Protein 1) and CTLA-4 (Cytotoxic T-Lymphocyte-Associated Antigen 4)-two key immune checkpoint receptors. It is designed as a novel tetrameric construct that preferentially binds to tumor-infiltrating lymphocytes (TILs) co-expressing PD-1 and CTLA-4 in the tumor microenvironment (withhigher avidity than in peripheral tissues).This study aims to investigate the therapeutic efficacy and safety of recombinant oncolytic adenovirus (KD01) in patients with gynecologic malignancies. Meanwhile, it will explore the impact of KD01 on the immune function of cervical cancer patients as well as its tumor cell-killing mechanism. This research is expected to provide novel strategies and approaches for the treatment of gynecologic malignancies, and contribute to improving the rehabilitation and quality of life of patients.

The study is divided into Phase I and Phase II. Phase II consists of Cohort A (cervical cancer cohort) and Cohort B (endometrial cancer cohort).Phase I will include patients with gynecologic malignancies who have failed systemic therapy.Phase II will include reproductive-aged women with a strong desire to preserve fertility.Phase II Cohort A will include patients with cervical squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma, staged as IB1 (tumor size ≥1 cm), IB2, IB3 (tumor size ≤5 cm) and IIA1 (based on FIGO 2018 staging system); baseline MRI examination confirms that the lesion does not involve the lower uterine segment; for patients in Stage II , the length of vaginal involvement is < 2 cm.Phase II Cohort B will include patients with endometrial atypical hyperplasia or endometrial adenocarcinoma (FIGO Grade 1-Grade 2, FIGO 2023 Stage IA1 and IA2), with mismatch repair deficiency (MMRd) or no response to progestogen therapy; baseline MRI examination combined with chest CT or PET/CT confirms that the lesion is limited to the endometrial layer or superficial myometrium, without obvious involvement of the deep myometrium, cervix or extrauterine sites.

ELIGIBILITY:
Inclusion Criteria -1.Phase I: Patients with gynecologic malignancies who have failed systemic therapy. Specifically, histologically or cytologically confirmed gynecologic malignancies that have progressed after adequate treatment and for which no effective therapy is available, or no standard therapy exists.Age: 18 to 75 years old (inclusive).

Phase II: Reproductive-aged women with a strong desire to preserve fertility, who understand and accept potential risks (recommended age ≤ 40 years old).Cohort A (Cervical Cancer Cohort): Histologically confirmed cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma, staged as IB1 (tumor size ≥ 1 cm), IB2, IB3 (tumor size ≤ 5 cm), or IIA1 (FIGO 2018 ). Baseline MRI confirms no involvement of the lower uterine segment; vaginal involvement length < 2 cm for Stage II patients.Cohort B (Endometrial Cancer Cohort): Histologically confirmed endometrial atypical hyperplasia or endometrial adenocarcinoma (FIGO Grade 1-Grade 2, FIGO 2023 Stage IA1 and IA2), with mismatch repair deficiency (MMRd) or no response to progestogen therapy. Baseline MRI combined with chest CT or PET/CT confirms lesions are limited to the endometrial layer or superficial myometrium, with no obvious involvement of the deep myometrium, cervix, or extrauterine sites.

* 2.Eastern Cooperative Oncology Group (ECOG) Performance Status: 0 or 1.
* 3.Expected Survival: ≥ 3 months.
* 4.No major organ dysfunction, including but not limited to hematopoietic, cardiac, pulmonary, hepatic, and renal function.

Hematological system ( no blood transfusion or hematopoietic stimulant therapy administered within 14 days prior to screening)：

1. Absolute Neutrophil Count (ANC)≥ 1.5 × 10⁹/L
2. Platelet Count (PLT)≥ 75 × 10⁹/L
3. Hemoglobin (Hb)≥ 90 g/L Hepatic System：

a.Total Bilirubin (TBIL)≤ 1.5 × Upper Limit of Normal (ULN) b.Alanine Aminotransferase (ALT)≤ 3 × ULN; ≤ 5 × ULN for patients with liver metastases or primary liver cancer c.Aspartate Aminotransferase (AST)≤ 3 × ULN; ≤ 5 × ULN for patients with liver metastases or primary liver cancer

Renal System:

1. Creatinine (Cr)≤ 1.5 × ULN
2. Creatinine Clearance (Ccr) (calculated only if Cr > 1.5 × ULN)> 50 mL/min (per Cockcroft-Gault formula)

Coagulation System:

1. Activated Partial Thromboplastin Time (APTT)≤ 1.5 × ULN
2. International Normalized Ratio (INR)≤ 1.5 × ULN

   * 5.Premenopausal female subjects must have a negative pregnancy test at screening.All subjects of childbearing potential must agree to use a reliable contraceptive method (barrier contraception or abstinence) with their partners from screening until at least 3 months after the last dose of study drug.
   * 6.Informed Consent: Voluntarily signs a written informed consent form prior to study participation, with a full understanding of the trial.

Exclusion Criteria

* 1.History of Severe Cardiovascular and Cerebrovascular Diseases, including but not limited to:

  1. Severe cardiac rhythm or conduction abnormalities requiring clinical intervention (e.g., symptomatic ventricular arrhythmias, Grade II-III atrioventricular block);
  2. Corrected QT interval (QTcF) ≥ 460 ms on 12-lead electrocardiogram at rest;
  3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade ≥ 3 cardiovascular events within 6 months prior to the first dose;
  4. New York Heart Association (NYHA) Functional Class ≥ II, left ventricular ejection fraction (LVEF) < 50%, or other structural heart diseases deemed high-risk by the investigator;
  5. Clinically uncontrolled hypertension.
* 2.Phase II: Imaging evidence of significant retroperitoneal lymph node metastasis;Cohort A (Cervical Cancer Cohort): Imaging evidence of lower uterine segment or endometrial involvement; Cohort B (Endometrial Cancer Cohort): Imaging evidence of deep myometrial, cervical, or extrauterine tumor invasion.
* 3.Clinically significant serous effusion requiring intervention within 4 weeks prior to informed consent.
* 4.History of autoimmune disease, immune system dysfunction, or organ transplantation.
* 5.Active infection requiring systemic anti-infective therapy (routine prophylactic anti-infective therapy per clinical trial institution is excluded); or unexplained fever > 38.5°C during screening.
* 6.Positive results for human immunodeficiency virus antibody (HIV-Ab) or treponema pallidum antibody; active hepatitis B (hepatitis B surface antigen [HBsAg] positive with HBV-DNA > 500 IU/mL or above the lower limit of detection of the clinical trial institution, if the lower limit is higher than 500 IU/mL); active hepatitis C (patients with positive HCV antibody but undetectable HCV-RNA are eligible). Patients receiving prophylactic antiviral therapy (excluding interferon) are eligible.
* 7.Uncontrolled seizures, central nervous system disorders, or psychiatric conditions resulting in cognitive impairment.
* 8.Adverse reactions from prior anti-tumor therapy have not resolved to grade ≤ 1 (per the Common Terminology Criteria for Adverse Events (CTCAE) v5.0), with the exception of toxicities judged by the investigator to pose no safety risks (e.g., alopecia).
* 9.Current requirement for antiviral therapy, or use of antiviral drugs within 2 weeks prior to the first dose of study drug.
* 10.Receipt of nitrosourea or mitomycin C within 6 weeks prior to the first dose;Receipt of oral fluoropyrimidines or small-molecule targeted agents within 2 weeks prior to the first dose or within 5 half-lives of the drug (whichever is longer);Receipt of traditional Chinese medicine with anti-tumor indications within 2 weeks prior to the first dose;Receipt of other chemotherapy, radiotherapy, biological therapy, endocrine therapy (excluding progestogen use in Phase II Cohort B), immunotherapy, etc., within 4 weeks prior to the first dose.
* 11.Receipt of systemic glucocorticoids (prednisone > 10 mg/day or equivalent dose of similar drugs) or other immunosuppressive agents within 14 days prior to the first dose, excluding: Topical, ophthalmic, intra-articular, intranasal, or inhaled glucocorticoid therapy;Short-term glucocorticoid use for prophylactic purposes (e.g., prevention of contrast-induced allergy).
* 12.Prior treatment with oncolytic viruses or oncolytic bacteria.
* 13.Vaccination within 28 days prior to the first dose.
* 14.Pregnant or lactating women.
* 15.History of severe allergies or allergic diathesis.
* 16.Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with cervical malignancies
Enrollment: 97 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
SAEs and AEs in Phase I | 2 years
  Incidence of serious adverse events (SAEs), incidence and severity of adverse events (AEs).
MTD and RD in Phase I | 2 years
  Determine the maximum tolerated dose (MTD) based on the incidence of dose-limiting toxicities (DLTs), and derive the recommended dose (RD) for monotherapy.
ORR in Phase II Cohort A | 2 years
  Objective response rate (ORR) following neoadjuvant therapy (preoperative treatment).
CR in Phase II Cohort B | 6 months
  Complete response (CR) rate at 6 months.

SECONDARY OUTCOMES:
Biodistribution in Phase I | 2 years
  The detected concentrations of KD01 in blood, urine, feces, saliva, and injection site tissues.
RFS in Phase II | 2 years
  2-year recurrence-free survival (RFS) rate.
pCR in Phase II Cohort A | 2 years
  Pathological complete response (pCR) rate following neoadjuvant therapy (preoperative treatment)
Disease response rate in Phase II Cohort B | 12 months
  Disease response rate at 12 months.
SAEs and AEs in Phase II | 2 years
  Incidence of serious adverse events (SAEs), incidence and severity of adverse events (AEs).

OTHER OUTCOMES:
Anti-Ad5 adenovirus antibody | 2 years
  Dynamic changes in anti-Ad5 adenovirus antibody titers.
Immunogenicity | 2 years
  Dynamic changes in ADA and NAb of KD01.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No